CLINICAL TRIAL: NCT06003153
Title: GLUCOSE-MGH: Genetic Links Understood Through Challenge With Oral Semaglutide Exposure at MGH
Acronym: GLUCOSE-MGH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Josephine Li, MD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023P001852; K23DK131345 (NIH)
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Genetic Predisposition; Metabolic Diseases; Type 2 Diabetes
MeSH Terms: conditions — Genetic Predisposition to Disease; Metabolic Diseases; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- GLUCOSE-MGH Study (Other): Day 1: Mixed meal tolerance test
  Day 3-15: 7 mg oral semaglutide, once daily
  Day 16: 1 dose of 7 mg oral semaglutide, Mixed meal tolerance test in the presence of semaglutide
  Interventions: Drug: oral semaglutide; Other: Mixed Meal Tolerance Test (MMTT)

INTERVENTIONS:
Drug: oral semaglutide — Semaglutide is the only oral glucagon-like peptide 1 receptor agonist (GLP-1 RA) approved for treatment of type 2 diabetes. Participants will receive 7 mg of oral semaglutide once daily for 14 days in between Visit 1 and Visit 2.
Other: Mixed Meal Tolerance Test (MMTT) — The MMTT is developed by the Metabolism and Nutrition Metabolic Kitchen at the MGH TCRC. The meal is a high-calorie, high-carbohydrate and moderate-to-high glycemic index challenge composed of commonly consumed breakfast food items. It provides nearly 90 grams of carbohydrates and mimics an oral glucose challenge. The participants will undergo a MMTT at Visit 1 and Visit 2.

SUMMARY:
The goal of this research study is to evaluate the pathophysiologic mechanisms by which genetic variation impacts response to an FDA-approved medication commonly used to treat type 2 diabetes called oral semaglutide (Rybelsus) and to characterize the physiological response to a mixed meal tolerance test (MMTT) before and after a 14-day treatment with oral semaglutide. The investigators will do this by measuring factors in the blood, such as sugars, fats, metabolites, and proteins, after eating a standardized breakfast meal at the first visit and after taking 14 doses of oral semaglutide over two weeks before the second study visit. The food (mixed meal breakfast) we will be studying is specially prepared to contain a set amount of protein, carbohydrates, and fat. The investigators hypothesize that understanding how the acute biochemical response to oral semaglutide differs by genetic variation will generate insight into drug mechanisms and type 2 diabetes pathophysiology.

DETAILED DESCRIPTION:
On day 1 (Visit 1), the research subject will present to the Translational and Clinical Research Center (TCRC) after an overnight fast. We will obtain informed consent, check vital signs, take anthropometric measurements, and draw fasting blood work through an intravenous catheter. The subject will then be provided a standard mixed meal to be consumed within 30 minutes. Additional blood will be drawn at the time of meal completion (0 minutes), as well as 5, 15, 30, 60, 90, and 120 minutes following the meal. During study days 3-15, the subject will take 7 mg of oral semaglutide once daily. On day 16 (Visit 2), the research subject will return to the TCRC. During this visit, the subject will take the final (14th) dose of semaglutide, receive fasting blood work, and receive another mixed meal with subsequent blood draws at several time points over 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females
2. Ages 18-50 (inclusive)
3. Able/willing to give consent
4. Span the metabolic range between normal glycemia and pre-diabetes (fasting glucose of 100-125 mg/dL based on chart review of existing laboratory data)

Exclusion Criteria:

1. Currently taking medications or intending to take medications for diabetes
2. Currently taking medications or intending to take medications that affect glycemic parameters, such as glucocorticoids, growth hormone, or fluoroquinolones
3. Personal history of intestinal malabsorption, bariatric surgery, celiac disease, gallbladder disease, or pancreatitis
4. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2
5. Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2 per the Modification of Diet in Renal Disease equation
6. History of cirrhosis and/or aspartate aminotransferase or alanine aminotransferase more than 3x upper limit of normal
7. Dietary restrictions preventing consumption of a MMTT
8. Women who are pregnant, nursing, or at risk of becoming pregnant
9. Participation in other interventional studies during the current study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Insulin response to oral semaglutide treatment | 15 days
  Investigators will measure the change in insulin area under the curve (AUC) over 120 minutes of the MMTT, calculated using the trapezoidal method, between Visit 1 and Visit 2 as an index of response to oral semaglutide, and compare this outcome by genotype at selected loci.

SECONDARY OUTCOMES:
Fasting glucose response to oral semaglutide treatment | 15 days
  Investigators will measure the change in fasting glucose over 120 minutes of the MMTT, between the two visits, and compare this outcome by genotype at selected loci.
Cumulative glucose response to oral semaglutide treatment | 15 days
  Investigators will measure the change in glucose area under the curve (AUC) over 120 minutes of the MMTT, between the two visits, and compare this outcome by genotype at selected loci.
Baseline incretin level | 120 minutes during Visit 1
  Investigators will measure levels of GLP-1 during the length of the baseline MMTT (120 minutes) that takes place on Visit 1, and compare changes in the baseline levels by genotype at selected loci.

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Li, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States